CLINICAL TRIAL: NCT05600413
Title: L-Citrulline Supplementation to Improve Vascular Function and Responsiveness at Rest and During Exercise in Postmenopausal Women
Brief Title: Citrulline Supplementation On Vascular Responsiveness and Function in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Arturo Figueroa, Principal Investigator, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB2019-1197
Record Dates: First submitted 2022-10-24; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Menopause
Keywords: Endothelial function; Blood pressure; Blood flow
MeSH Terms: interventions — Citrulline

STUDY DESIGN:
Intervention Model Description: Double (Participant, Investigator) Randomized, double-blind, placebo-controlled, parallel study design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Citrulline (Experimental): L-Citrulline: 6 grams/day
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Crystalline Cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — 4 weeks of L-Citrulline supplementation (6 grams/day)
  Arms: L-Citrulline
Dietary Supplement: Placebo — 4 weeks of Placebo (crystalline cellulose)
  Arms: Placebo

SUMMARY:
The objective of this project is to provide evidence that L-Citrulline (L-CIT) supplementation can improve vascular function at rest and in response to exercise in postmenopausal women.

DETAILED DESCRIPTION:
L-CIT is a non-essential amino acid that is a precursor to L-arginine, the substrate used to produce an important vasodilatory molecule called nitric oxide. The purpose of this study is to identify the effects of 6 grams of L-CIT for 4 weeks on vascular function (endothelial function, blood flow, muscle oxygenation, and blood pressure) at rest and in response to different stressors (cold pressor test, isometric and dynamic exercise).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (absence of menstruation > 1 year) between the ages of 50 - 79 years.
* Sedentary ( < 120 minutes of exercise/week)
* Resting systolic blood pressure < 150 mmHg and diastolic blood pressure < 90 mmHg
* Not participating as a subject in another study for at least 2 months prior to the study and for the duration of the study
* Willingness to abstain from food supplements 1 month prior to the start of the study and throughout the duration of the study

Exclusion Criteria:

* Body mass index ≥ 40
* Currently taking more than one vasoactive drug for blood pressure control
* Cardiometabolic diseases or other chronic diseases
* Taking hormone replacement therapy 3 months prior to the study
* Current or prior use of tobacco products
* More than a moderate intake of alcohol
* Use of medications and/or supplements that may affect outcome variables
* Musculoskeletal disorders that will prevent exercise performance

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Microvascular endothelial function | 4 weeks
  Endothelial function will be assessed via reactive hyperemic index using the EndoPAT device.
Changes in brachial and aortic blood pressure responses via automated sphygmomanometry during metaboreflex activation | 4 weeks
  Brachial and aortic blood pressures (systolic and diastolic) will be assessed using an arm cuff during isometric handgrip exercise and postexercise muscle ischemia.
Changes in aortic hemodynamics using pulse wave analysis during metaboreflex activation | 4 weeks
  The speed and reflection pressures, both representing aortic hemodynamic parameters, will be assessed using radial applanation tonometry and a validated transfer function (AtCor Medical) during isometric handgrip exercise and postexercise muscle ischemia.
Blood flow during dynamic exercise | 4 weeks
  Blood flow will be measured using ultrasound in the superficial femoral and brachial artery during dynamic exercises superimposed with the cold pressor test.
Muscle oxygenation during dynamic exercise | 4 weeks
  Muscle oxygenation will be measured using near infrared spectroscopy during dynamic exercises superimposed with the cold pressor test.

SECONDARY OUTCOMES:
Serum nitric oxide levels | 4 weeks
  Serum levels of nitric oxide will be assessed.
Changes in brachial and aortic blood pressure responses via automated sphygmomanometry during dynamic plantarflexion exercise and handgrip combined with the cold pressor test | 4 weeks
  Brachial and aortic blood pressures (systolic and diastolic) will be assessed using an arm cuff during dynamic plantarflexion exercise and handgrip combined with the cold pressor test.
Changes in aortic hemodynamics using pulse wave analysis during dynamic plantarflexion exercise and handgrip combined with the cold pressor test | 4 weeks
  The speed and reflection pressures, both representing aortic hemodynamic parameters, will be assessed using radial applanation tonometry and a validated transfer function (AtCor Medical) during dynamic plantarflexion exercise and handgrip combined with the cold pressor test.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Figueroa, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No